CLINICAL TRIAL: NCT03220958
Title: A Randomized Placebo Controlled Trial of IV Metoclopramide for Acute Post-traumatic Headache
Brief Title: Metoclopramide for Post Traumatic Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-7898
Record Dates: First submitted 2017-04-19; First posted 2017-07-18 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Metoclopramide; Diphenhydramine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metoclopramide (Experimental): Metoclopramide 20mg + diphenhydramine 25mg + 100cc normal saline, administered as an intravenous drip
  Interventions: Drug: Metoclopramide; Drug: Diphenhydramine; Drug: Normal saline
- Placebo (Placebo Comparator): Normal saline, administered as an intravenous drip
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Metoclopramide — Metoclopramide 20mg
  Arms: Metoclopramide
Drug: Diphenhydramine — Diphenhydramine 25mg
  Arms: Metoclopramide
Drug: Normal saline — 100ml normal saline

SUMMARY:
Nearly 1.5 million patients present to US emergency departments annually following head trauma. Headache is a frequent symptom of victims of head trauma. The purpose of this study is to see if an intravenous medication called metoclopramide can improve the symptoms of patients with acute post-traumatic headache.

ELIGIBILITY:
Inclusion Criteria:

Included patients will be adults who meet International Classification of Headache Disorders criteria for acute post-traumatic headache. These are as follows:

* Traumatic injury to the head has occurred
* Headache has developed within 7 days of injury to the head
* Headache is not better accounted for by another diagnosis (eg, previous history of migraine or tension-type headache)

The headache must be rated as moderate or severe in intensity at the time of initial evaluation.

Exclusion Criteria:

Patients will be excluded if more than ten days have elapsed since the head trauma, if the headache has already been treated with an anti-dopaminergic medication, or for medication contra-indications including pheochromocytoma, seizure disorder, Parkinson's disease, use of MAO inhibitors, and use of anti-rejection transplant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman BW, Irizarry E, Cain D, Caradonna A, Minen MT, Solorzano C, Zias E, Zybert D, McGregor M, Bijur PE, Gallagher EJ. Randomized Study of Metoclopramide Plus Diphenhydramine for Acute Posttraumatic Headache. Neurology. 2021 May 4;96(18):e2323-e2331. doi: 10.1212/WNL.0000000000011822. Epub 2021 Mar 24. PMID 33762421

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide | Placebo
Started | 81 | 79
Completed | 81 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide | Placebo | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (16) | 46 (17) | 45 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 56 | 107
  Male | 30 | 23 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160
Baseline pain intensity, as measured on a 0-10 scale [Mean (Standard Deviation); unit: units on a scale] | 8.3 (1.6) | 8.3 (1.5) | 8.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: 0-10 Pain Scale on Which 0 = no Pain and 10= the Worst Pain Imaginable
Description: Improvement in this 0 to 10 verbal rating scale
Time Frame: 1 hour after medication administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metoclopramide | Placebo
Number analyzed (Participants) | 81 | 79
units on a scale | 5.2 (2.3) | 3.8 (2.6)

2. Secondary Outcome: Sustained Headache Relief
Description: Achieving a headache intensity of mild or none in the ED without use of rescue medication and maintaining a level of mild or none. Participants rate their headache as none, mild, moderate, or severe
Time Frame: 48 hours after medication administration
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide | Placebo
Number analyzed (Participants) | 78 | 76
Participants | 24 | 18

3. Secondary Outcome: Headache Days
Description: Number of days with any headache. Participants report the actual number of days they experienced headache. A "day" begins when they awake for the beginning of daily activities and ends when they go to sleep after completion of daily activities
Time Frame: 7 days after ED visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Metoclopramide | Placebo
Number analyzed (Participants) | 76 | 71
days | 3.3 (1.6) | 3.3 (1.6)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Metoclopramide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 35/81 | 22/79
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide (N=81) | Placebo (N=79)
Drowsiness (Nervous system disorders) | 15 (15) | 8 (8)
Akathisia (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Post-concussive syndrome (Nervous system disorders) | 7 | 5
Various other (Investigations) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03220958/Prot_SAP_002.pdf